CLINICAL TRIAL: NCT06696131
Title: Tenecteplase (TNK) in the Treatment of Intracerebral Hemorrhage (ICH)
Acronym: TNK in ICH
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gaurav Gupta, MD (Other)
Responsible Party: Sponsor-Investigator, Gaurav Gupta, MD, Principal Investigator; Professor | Department of Neurosurgery, RWJMS System Co-Director, Cerebrovascular & Endovascular Neurosurgery, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2024001604
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Intracerebral Hemorrhage; Intracranial Hemorrhages; Hemorrhagic Strokes
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TNK (Experimental): Participants would be given TNK through a brain catheter to dissolve an intracerebral blood clot after a hemorrhage.
  Interventions: Drug: TNK

INTERVENTIONS:
Drug: TNK — TNK will be delivered into the site of the intracerebral hemorrhage via a brain catheter.

SUMMARY:
The overall purpose of this study is to look at the safety and effectiveness of administering Tenecteplase (TNK) into the brain bleed (hematoma) instead of another clot-dissolving drug known as recombinant tissue plasminogen activator (rtPA), which is the current standard practice. Clot dissolving (Fibrinolytic) drugs work to break down blood clots and have been found to improve health outcomes when applied directly into the hematoma within the brain. Patients who take part in this study will undergo the same surgical procedure that would normally be performed to treat them, but with the exception of TNK not rtPA.

ELIGIBILITY:
Inclusion Criteria

* Patient/legally authorized representative has signed the Informed Consent Form.
* Ability to comply with the study protocol, in the investigator's judgment.
* Patients 18 to 80 years of age with an ICH had occurred within 24 hours before admission.
* Spontaneous supratentorial (basal ganglia, thalamus, lobar) ICH ≥30 mL measured utilizing the ABC/2 method.
* Subjects with a GCS score of 5-14.
* NIHSS ≥6.
* Stability CT scan done at least 6 hours after baseline CT showing clot stability (growth <5 mL as measured by ABC/2 method). If the hematoma volume measured on the stability CT scan increases by 5 mL or more, a second stability CT scan will be performed 12 hours later.
* Sustained systolic blood pressure (SBP) <180 mm Hg for six hours recorded closest to the time of drug administration.
* Symptoms must be present less than 24 hours prior to baseline CT scan.
* Baseline Rankin score of 0 or 1.

Exclusion Criteria

* Presence of infratentorial parenchymal bleeding.
* Presence of a hemorrhage extending to the midbrain.
* An unknown time of onset or the symptoms onset more than 24 hours prior to admission.
* Pregnancy.
* Inability to obtain written informed consent from subject or legal representative.
* Sustained SBP >180 mm Hg for six hours recorded closest to the time of drug administration.
* Age <18 and >80 years.
* Radiological evidence of arterio-venous malformation, aneurysm, amyloid angiopathy, Moyamoya disease, hemorrhagic conversion of an ischemic stroke, recurrent hemorrhage in the same location within the past 365 year or unstable mass as a source for the ICH.
* Evidence of coagulopathy (international normalized ratio >1.3; platelet count <100 ,000 or platelet dysfunction P2Y-12 >250) or known clotting disorder.
* Bilateral fixed, dilated pupils indicating irreversible impaired brain stem function with GCS ≤4.
* Patients with severe ICH and IVH who require an external ventricular drain (EVD) placement for cerebrospinal fluid (CSF) diversion or separate intraventricular thrombolysis.
* Inability to maintain INR less than 1.3.
* Use of anticoagulants prior to symptom onset and subjects requiring long-term anticoagulants (the reversal is permitted if the patient can tolerate the short-term risk of reversal).
* Use of Dabigatran, Apixaban, and/or Rivaroxaban (or a similar medication from the similar medication class) prior to symptom onset.
* Internal bleeding (GI, renal, respiratory etc).
* Mechanical heart valve (Bioprosthetic heart valve is permitted).
* Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis (atrial fibrillation without mitral stenosis is permitted).
* Allergy or sensitivity to TNKase.
* Participation in a concurrent clinical trial.
* Serious illness (advanced stage which can interfere with the outcome).
* The patient is unstable and would not benefit from a surgical intervention.
* GCS score of 3-4 and 15 (to ensure patient safety and study feasibility).
* Historical mRS score of 2-6 (at admission).
* Symptomatic tract hemorrhage or a tract hemorrhage more than 5 mm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | From treatment until follow-up date (+/- 30 days)
  To assess the safety of 0.25 mg TNKase (single dose) administered directly into the hematoma via a soft brain catheter in patients with ICH.
Adverse Event Evaluation | From treatment until follow-up date (+/- 30 days)
  To evaluate the incidence and severity of adverse events, such as rehemorrhage, infection, mortality at 30 days following the administration of TNKase.

SECONDARY OUTCOMES:
Radiological Assessment of the Hematoma Resolution | From treatment until follow-up date (+/- 30 days)
  Using radiological imaging, we will assess the resolution of the hematoma from the brain with the end of treatment volume goal as 15 ml and compare these findings to baseline imaging obtained prior to TNKase administration

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — Rutgers University, RWJ Medical School

IPD SHARING:
Plan to Share IPD: No